CLINICAL TRIAL: NCT03456297
Title: Web-based Clinical Pedagogy Program to Enhance Nurse Preceptors' Teaching Competency and Nursing Students' Learning Outcomes in Clinical Competency
Brief Title: Web-based Clinical Pedagogy Program to Enhance Nurse Preceptors' Teaching Competency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Vivien Xi WU, PhD, Lecturer, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MOE2017-TRF-009
Record Dates: First submitted 2018-02-20; First posted 2018-03-07 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Web-based Program for Nurse Preceptors
Keywords: Web-based clinical pedagogy program; nurse preceptors; teaching competency

STUDY DESIGN:
Intervention Model Description: A prospective cluster randomisation trial will be used for this study. The Web-based Clinical Pedagogy Program will be provided to the participants in the experimental cluster, while the participants in the control cluster will receive the current preceptorship course.
Who Masked: Participant
Masking Description: The 10 clinical departments will be randomised into two clusters, experimental and controlled clusters. The participants will be randomised based on the department that they work in. The advantage of the cluster randomised controlled trial is the ability to control for "contamination" across individuals, for example, one individual's use of WCP may influence another individual in the same department (Kellar & Kelvin, 2013).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental cluster (Experimental): The Web-based clinical pedagogy program (WCP) will be provided to the participants in the experimental cluster.
  Interventions: Other: Web-based clinical pedagogy program (WCP)
- Control cluster (No Intervention): The participants in the control cluster will receive the current face-to-face preceptorship course.

INTERVENTIONS:
Other: Web-based clinical pedagogy program (WCP) — The nurse preceptors in the experimental cluster will be given access to download the WCP on mobile devices. The unique interactive features provide continuous support and allow preceptors to discuss the clinical encounters with their peers and consult experts for advice.
  Arms: Experimental cluster

SUMMARY:
The study aims to develop a Web-based clinical pedagogy program (WCP) for nurse preceptors; compare the WCP with the current preceptorship course on clinical teaching competence, assessment techniques and self-efficacy; examine nurse preceptors' attitudes toward Web-based learning; and explore the preceptors' perspectives of WCP.

DETAILED DESCRIPTION:
Clinical nursing education provides opportunities for students to learn in multiple patient care settings, receive appropriate guidance, and foster the development of clinical competence and professionalism. Nurse preceptors guide students to integrate theory into practice, teach clinical skills, assess clinical competency, and enhance problem solving and critical thinking skills. Previous researches have indicated that the teaching competency of the nurse preceptors can be transferred to the students' clinical learning to enhance their clinical competencies. Web-based learning is recognised as an effective learning approach for enhancing nursing knowledge and skills. The flexible and resource-rich nature of Web-based learning may encourage nurses to use it as a platform for continuing education.

The present study aims to develop a Web-based clinical pedagogy program (WCP) for nurse preceptors; compare the WCP with the current preceptorship course on clinical teaching competence, assessment techniques and self-efficacy; examine nurse preceptors' attitudes toward Web-based learning, and explore the preceptors' perspectives of WCP .

The design of the components in WCP is grounded on Bandura's self-efficacy theory. The WCP is an evidence-based program which provides a comprehensive coverage on clinical teaching pedagogy and assessment strategies. The unique web-based technology and interactive features provide a platform to allow the nurse preceptors to discuss the clinical encounters with their peers, and consult the experts. The WCP provides flexibility in learning, which may match the tight work schedule of the preceptors and aligns with the initiative of Singapore government to encourage leveraging on technology and continuing education for citizens.

A prospective cluster randomisation trial will be used for this study. The WCP will be provided to the preceptors in the experimental cluster, while the preceptors in the controlled cluster will receive the current preceptorship course. A follow-up qualitative study using focus group will be conducted to further explore the preceptors' perspectives of WCP.

Clinical teaching competence inventory (CTCI), preceptor self-efficacy assessment instrument (PSAI), attitudes towards web-based continuing learning survey (AWCLS) will be used to evaluate preceptors' learning outcomes. Socio-demographic data will be collected for both groups at baseline. Nurse preceptors will be invited to complete questionnaires on CTCI, PSAI, and AWCLS at three time points, before the learning program (baseline), after the learning program (post-test 1), and after clinical teaching experience (post-test 2). In addition, 16 preceptors will be invited to participate in the focus group discussions.

Ministry of Health, Singapore encourages strategies that are innovative and promote professional development of healthcare professionals, who feel more motivated and dignified to care for the health of the population. It is paramount that continuing education courses integrate with technology, increase the flexibility and responsiveness of the nursing workforce, and offer alternative means to take up courses.

ELIGIBILITY:
Inclusion Criteria:

* nurse preceptors and clinical nurse leaders;
* guiding the nursing students for clinical teaching and assessment;
* 21 years old and above;
* have not completed the clinical teaching course provided by the hospital; and
* possess and able to use smart mobile devices (Smart phone, tablet, or laptop) in daily lives.

Exclusion Criteria:

* nurse preceptors who do not know how to use the smart mobile devices.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Preceptor Self-efficacy Questionnaire (PSEQ) | Change from Baseline PSEQ at 6 months
  The PSEQ (Parsons, 2007) consists of 21 items, and assesses the confidence in preceptor skills using a four-point Likert scale

SECONDARY OUTCOMES:
Clinical Teaching Competence Inventory (CTCI) | Change from Baseline CTCI at 6 months
  The CTCI consists of four domains of teaching and assessment competencies and 31 items on a five-point Likert scale. The four domains are: student evaluation (assessment), goal setting and individual teaching, teaching strategies, and demonstration of organized knowledge.
Attitudes toward Web-based Continuing Learning Survey (AWCLS) | Change from Baseline AWCLS at 6 months
  There are four dimensions and 18 items using a 7-point Likert scale in the survey. The four dimensions are the perceived usefulness scale assesses the nurses' perceptions of the extent to which they perceive that the influence of web-based continuing learning is useful; the perceived ease of use scale evaluates the nurses' perceptions of the extent to which web-based continuing learning is easy to use; the behaviour scale measures the nurses' willingness to take up web-based continuing learning; and the affection scale assesses the nurses' perceptions regarding positive feelings about web-based continuing learning.

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Xi Wu, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
study protocol and final report will be submitted to peer-reviewed journal for possible publication.

REFERENCES:
- [Background] Wu XV, Chan YS, Tan KHS, Wang W. A systematic review of online learning programs for nurse preceptors. Nurse Educ Today. 2018 Jan;60:11-22. doi: 10.1016/j.nedt.2017.09.010. Epub 2017 Sep 28. PMID 28987893
- [Background] Wu XV, Enskar K, Pua LH, Heng DGN, Wang W. Clinical nurse leaders' and academics' perspectives in clinical assessment of final-year nursing students: A qualitative study. Nurs Health Sci. 2017 Sep;19(3):287-293. doi: 10.1111/nhs.12342. Epub 2017 Mar 30. PMID 28371304
- [Background] Wu XV, Enskar K, Heng DG, Pua LH, Wang W. The perspectives of preceptors regarding clinical assessment for undergraduate nursing students. Int Nurs Rev. 2016 Sep;63(3):473-81. doi: 10.1111/inr.12272. Epub 2016 Apr 21. PMID 27100137
- [Background] Wu XV, Wang W, Pua LH, Heng DG, Enskar K. Undergraduate nursing students' perspectives on clinical assessment at transition to practice. Contemp Nurse. 2015 Oct-Dec;51(2-3):272-85. doi: 10.1080/10376178.2016.1163232. Epub 2016 Mar 30. PMID 26956057